CLINICAL TRIAL: NCT00849914
Title: Expression Levels of microRNA Processing Enzymes Dicer and Drosha in Epithelial Skin Cancer
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: 005
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Punch biopsy from tumour, punch biopsy from healthy skin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with actinic keratoses of the skin
- 2: Patients with basal cell carcinoma of the skin
- 3: Patients with squamous cell carcinoma of the skin

SUMMARY:
MicroRNAs (miRNAs) are very small endogenous RNA molecules about 22-25 nucleotides in length, capable of post-transcriptional gene regulation. miRNAs bind to their target messenger RNAs (mRNAs), leading to cleavage or suppression of target mRNA translation based on the degree of complementarity. miRNAs have recently been shown to play pivotal roles in diverse developmental and cellular processes and linked to a variety of skin diseases and cancers. In the present study the expression profiles for the two most important miRNA processing enzymes Dicer and Drosha of actinic keratoses, basal cell carcinoma and squamous cell carcinoma are compared to healthy skin tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with actinic keratoses, squamous cell carcinoma or basal cell carcinoma of the skin

Exclusion Criteria:

* Patients under 18 years of age
* Patients with other forms of cancer in previous medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dermatologic primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Peter Altmeyer, Principal Investigator — Department of Dermatology and Allergology, Ruhr-University Bochum
Locations (1):
- Department of Dermatology and Allergology, Ruhr-University Bochum, Bochum, Germany

REFERENCES:
- [Result] Sand M, Gambichler T, Skrygan M, Sand D, Scola N, Altmeyer P, Bechara FG. Expression levels of the microRNA processing enzymes Drosha and dicer in epithelial skin cancer. Cancer Invest. 2010 Jul;28(6):649-53. doi: 10.3109/07357901003630918. PMID 20210522